CLINICAL TRIAL: NCT07053475
Title: IRONICA: IRON Repletion in Congestive Heart Failure - A Randomized Controlled Trial Comparing Oral Versus IV Approaches
Brief Title: IRONICA: IRON Repletion In Heart Failure - A Comparison of Oral and IV Approaches
Acronym: IRONICA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Syed Hamza Mufarrih (Other)
Collaborators: American Regent, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Syed Hamza Mufarrih, Principal Investigator, Western Kentucky Heart and Lung Research Foundation and Educational Trust
Organization: Western Kentucky Heart and Lung Research Foundation and Educational Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-11-18-Mufa-OralvsIV-Iron; AR2059 (Other Grant/Funding Number: American Regent, Inc.)
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction (HFrEF); Heart Failure With Preserved Ejection Fraction (HFPEF); Iron Deficiency; Iron-deficiency Anemia (IDA)
Keywords: Intravenous iron; Oral iron; Ferric carboxymaltose; Ferrous sulfate; Transferrin saturation (TSAT); Functional iron deficiency; 6-minute walk test (6MWT); Kansas City Cardiomyopathy Questionnaire (KCCQ); Quality of life; Randomized controlled trial; Congestive heart failure; HFpEF; HFrEF
MeSH Terms: conditions — Heart Failure; Iron Deficiencies; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Fosfomycin; ferryl iron; ferrous sulfate; Iron

STUDY DESIGN:
Intervention Model Description: Randomized, 1:1, parallel-group, open-label PROBE design comparing IV ferric carboxymaltose with oral ferrous sulfate in adults with heart failure and TSAT < 20 %.
Who Masked: Outcomes Assessor
Masking Description: Investigators and participants know group assignment. 6-minute walk test staff, data analysts, and clinical endpoint adjudicators remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV Iron (Ferric Carboxymaltose) (Experimental): Patients randomized to receive intravenous ferric carboxymaltose. Dosing includes a 1-gram IV infusion during the index hospital stay, followed by a second infusion at Week 6 (1,000 mg if > 70 kg or 500 mg if ≤ 70 kg).
  Interventions: Drug: Ferric Carboxymaltose
- Oral Iron (Ferrous Sulfate) (Active Comparator): Patients randomized to receive one capsule of oral ferrous sulfate (Ferrex 150 mg) every 48 hours for 12 weeks.
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Ferric Carboxymaltose — Intravenous infusion of 1 gram FCM during index hospital stay, followed by a second dose at Week 6 (1,000 mg if > 70 kg or 500 mg if ≤ 70 kg).
  Other Names: FCM, IV Iron
  Arms: IV Iron (Ferric Carboxymaltose)
Drug: Ferrous Sulfate — Oral administration of one 150 mg capsule every 48 hours for 12 weeks.
  Other Names: Ferrex, Oral Iron
  Arms: Oral Iron (Ferrous Sulfate)

SUMMARY:
The goal of this clinical trial is to learn which iron treatment works better for adults with congestive heart failure and low iron levels: intravenous (IV) iron given through a vein or oral (PO) iron taken by mouth. Participants must have heart failure with reduced ejection fraction (HFrEF) or preserved ejection fraction (HFpEF) and a transferrin-saturation (TSAT) level below 20 percent.

The main questions the study will answer are:

1. Does IV iron raise walking distance on a 6-minute walk test more than oral iron after 24 weeks?
2. Does IV iron improve symptoms and quality of life more than oral iron?
3. How do the two treatments compare for safety, side effects, and hospital readmissions/ mortality?

Researchers will compare IV ferric carboxymaltose with oral ferrous sulfate to see which option helps people feel and function better.

What participants will do

* Be randomly assigned by (like flipping a coin) to IV iron or oral iron.
* Receive either a one-time IV iron infusion (with possible repeat at 12 weeks) or take iron pills twice each day for 24 weeks.
* Visit the infusion clinic at 6 weeks for second dose of IV iron if needed.
* Visit the clinic at 12 weeks for a follow-up to gather follow-up data including

  1. A 6-minute walk test
  2. Brief symptom and quality-of-life surveys
  3. Blood tests to measure serum iron, ferritin, and transferrin saturation

This study will help doctors decide whether IV or oral iron is the safer, more effective way to treat iron deficiency in people with heart failure in our local community.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* BMI ≥18.0 kg/m²
* Hemoglobin:

> 9 g/dL and <14 g/dL for men > 9 g/dL and <13 g/dL for women

* Diagnosed with Congestive Heart failure:

HFrEF: EF ≤40% in any recent echocardiogram HFpEF: EF ≥50-55% without any prior EF ≤40%, and evidence of diastolic dysfunction per ASE/EACVI 2023 criteria-defined as either grade ≥2 or ≥2 supporting echo parameters (septal e' <7 cm/sec or lateral e' <10 cm/sec, E/e' ≥15, TR velocity >2.8 m/s, LA volume index ≥34 mL/m², LV septal or posterior wall thickness ≥1.2 cm, or LA area ≥20 cm² / diameter ≥3.8 cm.

* Documented elevated NT-proBNP based on BMI and rhythm:

BMI <35: ≥220 pg/mL (NSR) or ≥660 pg/mL (A-Fib) BMI ≥35: ≥125 pg/mL (NSR) or ≥375 pg/mL (A-Fib)

* NYHA Class II-IV
* Transferrin saturation (TSAT) <20%
* Hemoglobin <14 g/dL for men, < 13 g/dL for women.
* Stable on heart failure therapy for ≥2-4 weeks
* Currently prescribed a diuretic at home
* Ambulatory (able to walk >20 ft with minimal assistance)
* Willing and able to give informed consent

Exclusion Criteria:

* Received IV iron, ESA, or blood transfusion within the last 6-12 months
* Received high-dose oral iron (>100 mg/day in past 7 days)
* Severe renal impairment (eGFR <15 mL/min/1.73 m² or on dialysis)
* Patients with known cirrhosis or transaminitis with AST >141 or ALT >112 IU/L
* Active bleeding or known bleeding disorder
* Recent cardiac surgery, myocardial infarction, or stroke within past 3 months
* Active infection, defined as any systemic or deep-seated infection (e.g., bacteremia, sepsis, osteomyelitis, or infections requiring IV antibiotics or hospitalization) at the time of screening.
* Active malignancy or undergoing chemotherapy/radiotherapy
* Vitamin B12 or folate deficiency (unless corrected prior to enrollment)
* Chronic liver disease (with LFTs >3× upper limit of normal)
* Pregnant or breastfeeding women or those not using effective contraception
* Lacks capacity to consent or unable to comply with study procedures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in 6-Minute Walk Distance | Baseline and 12 weeks
  Change in distance (in meters) walked during the 6-minute walk test from baseline to 12 weeks.

SECONDARY OUTCOMES:
Change in NYHA Functional Class | Baseline and 12 weeks
  Change in New York Heart Association (NYHA) class from baseline to 12 weeks.
Change in Quality of Life | Baseline and 12 weeks
  Change in patient-reported quality of life scores as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
Change in Iron Stores | Baseline and 12 weeks
  Change in iron parameters including serum ferritin, serum iron, and transferrin saturation from baseline to 12 weeks.
All-Cause Mortality | Through 12 weeks
  Death from any cause during the 12-week study period.
Heart Failure Readmissions | Through 12 weeks
  Number of heart failure-related hospital readmissions within 12 weeks.
Major Adverse Cardiac Events (MACE) | Through 12 weeks
  Composite of cardiovascular death, myocardial infarction, or stroke during the 12-week study period.
Adverse Events Related to Study Drug | Through 12 weeks
  Frequency of reported adverse effects attributed to either ferric carboxymaltose or oral ferrous sulfate during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- The Medical Center, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) will be made available to researchers upon reasonable request, following publication of primary results. Data sharing will require a data use agreement and IRB approval.

REFERENCES:
- [Background] von Haehling S, Doehner W, Evertz R, Garfias-Veitl T, Derad C, Diek M, Karakas M, Birkemeyer R, Fillippatos G, Lainscak M, Butler J, Ponikowski P, Bohm M, Friede T, Anker SD. Ferric carboxymaltose and exercise capacity in heart failure with preserved ejection fraction and iron deficiency: the FAIR-HFpEF trial. Eur Heart J. 2024 Oct 5;45(37):3789-3800. doi: 10.1093/eurheartj/ehae479. PMID 39185895
- [Background] Alcaide-Aldeano A, Garay A, Alcoberro L, Jimenez-Marrero S, Yun S, Tajes M, Garcia-Romero E, Diez-Lopez C, Gonzalez-Costello J, Mateus-Porta G, Cainzos-Achirica M, Enjuanes C, Comin-Colet J, Moliner P. Iron Deficiency: Impact on Functional Capacity and Quality of Life in Heart Failure with Preserved Ejection Fraction. J Clin Med. 2020 Apr 22;9(4):1199. doi: 10.3390/jcm9041199. PMID 32331365
- [Background] Bekfani T, Pellicori P, Morris D, Ebner N, Valentova M, Sandek A, Doehner W, Cleland JG, Lainscak M, Schulze PC, Anker SD, von Haehling S. Iron deficiency in patients with heart failure with preserved ejection fraction and its association with reduced exercise capacity, muscle strength and quality of life. Clin Res Cardiol. 2019 Feb;108(2):203-211. doi: 10.1007/s00392-018-1344-x. Epub 2018 Jul 26. PMID 30051186
- [Background] Cleland JGF, Pellicori P, Graham FJ, Lane R, Petrie MC, Ahmed F, Squire IB, Ludman A, Japp A, Al-Mohammad A, Clark AL, Szwejkowski B, Critoph C, Chong V, Schiff R, Nageh T, Glover J, McMurray JJV, Thomson EA, Robertson M, Ford I, Kalra PA, Kalra PR; IRONMAN Study Group. Adjudication of Hospitalizations and Deaths in the IRONMAN Trial of Intravenous Iron for Heart Failure. J Am Coll Cardiol. 2024 Oct 29;84(18):1704-1717. doi: 10.1016/j.jacc.2024.08.052. PMID 39443013
- [Background] Manceau H, Ausseil J, Masson D, Feugeas JP, Sablonniere B, Guieu R, Puy H, Peoc'h K. Neglected Comorbidity of Chronic Heart Failure: Iron Deficiency. Nutrients. 2022 Aug 5;14(15):3214. doi: 10.3390/nu14153214. PMID 35956390
- [Background] Zhou X, Xu W, Xu Y, Qian Z. Iron Supplementation Improves Cardiovascular Outcomes in Patients with Heart Failure. Am J Med. 2019 Aug;132(8):955-963. doi: 10.1016/j.amjmed.2019.02.018. Epub 2019 Mar 7. PMID 30853478
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499